CLINICAL TRIAL: NCT04094532
Title: Ultrasound Guided Transversus Thoracic Muscle Plane Block for Open Heart Surgery: Randomized Controlled Double Blind Study
Brief Title: Transversus Thoracic Muscle Plane Block for Open Heart Surgery
Acronym: TTMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIACARDIAC
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Pain, Acute; Pain, Chest
MeSH Terms: conditions — Acute Pain; Chest Pain | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided transverse thoracic muscle plane block (Active Comparator)
  Interventions: Drug: Bupivacaine
- ultrasound guided sham block (Sham Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — Ultrasound guided 20 ml % 0.250 bupivacaine injection to transverse thoracic muscle plane bilaterally
  Arms: ultrasound guided transverse thoracic muscle plane block
Drug: Saline — Ultrasound guided 20 ml % 0.9 saline injection to transverse thoracic muscle plane bilaterally
  Arms: ultrasound guided sham block

SUMMARY:
Poststernotomy pain is a complication of cardiac surgery. Poorly controlled pain is associated with myocardial ischemia, cardiac arrhythmias, hypercoagulability, pulmonary complications, and increased rates of delirium and wound infection.

The transverse thoracic muscle plane (TTMP) block is a novel plane block that provide pain for sternotomy. The aim of this study was to evaluate the analgesic effect of ultrasound guided TTMP block in patients undergoing open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologist's physiologic state I-III patients Undergoing Open Heart Surgery

Exclusion Criteria:

chronic pain bleeding disorders renal or hepatic insufficiency patients on chronic non-steroidal anti-inflammatory medications emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | first 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postextubation 0-24 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murata H, Hida K, Hara T. Transverse Thoracic Muscle Plane Block: Tricks and Tips to Accomplish the Block. Reg Anesth Pain Med. 2016 May-Jun;41(3):411-2. doi: 10.1097/AAP.0000000000000374. No abstract available. PMID 27093277